CLINICAL TRIAL: NCT03661567
Title: A Prospective, Randomized, Controlled Phase Ⅱ Study of Preventively Use of Methylprednisolone After Split-course Chemoradiotherapy to Reduce the Risk of Radiation-induced Pulmonary Injury For Bulky Local Advanced None-small Cell Lung Cancer
Brief Title: Methylprednisolone After Split-course Chemoradiotherapy For Bulky Local Advanced None-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GASTO-1044
Record Dates: First submitted 2018-09-01; First posted 2018-09-07 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: methylprednisolone; Split-course Chemoradiotherapy; Radiation-induced Pulmonary Injury
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone (Experimental): Patients were treated with methylprednisolone after the first course of chest radiation and concurrent chemotherapy, once a day, 32 milligram (mg) for 7 days, 24 mg for the next 7 days, then 16mg for 7 days, and 8 mg for the last 7 days.
  Interventions: Radiation: chest radiation; Drug: concurrent chemotherapy; Drug: Methylprednisolone
- Observation (Active Comparator): Observation after the first course of chest radiation, methylprednisolone can only be used for therapeutic purpose in the presence of grade≥2 radiation induced lung injury(NCI-CTC4.0).
  Interventions: Radiation: chest radiation; Drug: concurrent chemotherapy

INTERVENTIONS:
Radiation: chest radiation — split-course chest radiation
Drug: concurrent chemotherapy — weekly docetaxel(25mg/㎡) and nedaplatin(25mg/㎡) concurrent with chest radiation
Drug: Methylprednisolone — Methylprednisolone after the first course of radiation, once a day, 32 milligram (mg) for 7 days, 24 mg for the next 7 days, then 16mg for 7 days, and 8 mg for the last 7 days.
  Arms: Methylprednisolone

SUMMARY:
This Phase II randomized controlled study is to determine the efficacy of the preventively use of methylprednisolone after split-course chemoradiotherapy (CCRT) in locally advanced non-small cell lung cancer with bulky tumor.

DETAILED DESCRIPTION:
This study is to determine the efficacy of the preventively use of methylprednisolone after split-course chemoradiotherapy(CCRT) in locally advanced non-small cell lung cancer with bulky tumor.

All patients received four cycles of weekly docetaxel (25mg/㎡) and nedaplatin (25mg/㎡)(DP), each of 1 day's duration, combined with split-course thoracic radiotherapy, with one-month break. In the experimental arm, patients were treated with methylprednisolone after the first course of radiation, once a day, 32 milligram (mg) for 7 days, 24 mg for the next 7 days,then 16mg for 7 days, and 8 mg for the last 7 days. Toxicities will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v. 4.0.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of NSCLC.
* Patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

  * Unresectable phase IIIA(N2) and IIIB lung cancer confirmed by PET/CT, CT or MRI.
  * Whole lung V20>=35% when giving 60Gy which is the minimum dose of radical irradiation.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Previously treated with chemotherapy or treatment-naive
* No previous chest radiotherapy, immunotherapy or biotherapy
* Hemoglobin≥10 mg/dL, platelet≥100000/μL,absolute neutrophil count ≥1500/μL
* Serum creatinine ≤1.25 times the upper normal limit(UNL), or creatinine clearance≥60 ml/min
* Bilirubin ≤1.5 times UNL, AST（SGOT）≤2.5 times UNL ,ALT（SGPT）≤2.5 times UNL,alkaline phosphatase ≤5 times UNL
* FEV1 >0.8 L
* CB6 within normal limits
* patients and their family signed the informed consents

Exclusion Criteria:

* Previous or recent another malignancy, except nonmelanoma skin cancer or cervical cancer in situ
* Contraindication for chemotherapy
* Malignant pleural or pericardial effusion.
* Women in pregnancy, lactation period, or no pregnancy test 14 days before the first dose
* Women who has the probability of pregnancy without contraception
* Tendency of hemorrhage
* In other clinical trials within 30 days
* Addicted in drugs or alcohol, AIDS patients
* Uncontrollable seizure or psychotic patients without self-control ability
* Severe allergy or idiosyncrasy
* Not suitable for this study judged by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
rate of grade≥2 radiation pneumonia(NCI-CTC4.0) | 1 year from the end of radiotherapy
  radiation-induced pulmonary injury is classified into 1-5 grades according to NCI-CTC4.0. The incidence of symptomatic radiation-induced pulmonary injury: the ratio of grade 2 and above radiation-induced pulmonary injury cases in 1 year after radio therapy to all cases can be evaluated .

SECONDARY OUTCOMES:
the rate of grade≥2 pulmonary ventilation and diffusion capacity decline | 1 year from the end of radiotherapy
  It is divided into grade 1-4 according to SOMA.
the rate of grade≥2 visible change in CT after radiation | 1 year from the end of radiotherapy
  It is divided into grade 1-4 according to SOMA.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Giridhar P, Mallick S, Rath GK, Julka PK. Radiation induced lung injury: prediction, assessment and management. Asian Pac J Cancer Prev. 2015;16(7):2613-7. doi: 10.7314/apjcp.2015.16.7.2613. PMID 25854336
- [Background] Marks LB, Bentzen SM, Deasy JO, Kong FM, Bradley JD, Vogelius IS, El Naqa I, Hubbs JL, Lebesque JV, Timmerman RD, Martel MK, Jackson A. Radiation dose-volume effects in the lung. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S70-6. doi: 10.1016/j.ijrobp.2009.06.091. PMID 20171521
- [Background] Barthelemy-Brichant N, Bosquee L, Cataldo D, Corhay JL, Gustin M, Seidel L, Thiry A, Ghaye B, Nizet M, Albert A, Deneufbourg JM, Bartsch P, Nusgens B. Increased IL-6 and TGF-beta1 concentrations in bronchoalveolar lavage fluid associated with thoracic radiotherapy. Int J Radiat Oncol Biol Phys. 2004 Mar 1;58(3):758-67. doi: 10.1016/S0360-3016(03)01614-6. PMID 14967431
- [Background] Trott KR, Herrmann T, Kasper M. Target cells in radiation pneumopathy. Int J Radiat Oncol Biol Phys. 2004 Feb 1;58(2):463-9. doi: 10.1016/j.ijrobp.2003.09.045. PMID 14751516
- [Background] Roberts CM, Foulcher E, Zaunders JJ, Bryant DH, Freund J, Cairns D, Penny R, Morgan GW, Breit SN. Radiation pneumonitis: a possible lymphocyte-mediated hypersensitivity reaction. Ann Intern Med. 1993 May 1;118(9):696-700. doi: 10.7326/0003-4819-118-9-199305010-00006. PMID 8460855
- [Background] Kainthola A, Haritwal T, Tiwari M, Gupta N, Parvez S, Tiwari M, Prakash H, Agrawala PK. Immunological Aspect of Radiation-Induced Pneumonitis, Current Treatment Strategies, and Future Prospects. Front Immunol. 2017 May 2;8:506. doi: 10.3389/fimmu.2017.00506. eCollection 2017. PMID 28512460
- [Background] Murshed H, Liu HH, Liao Z, Barker JL, Wang X, Tucker SL, Chandra A, Guerrero T, Stevens C, Chang JY, Jeter M, Cox JD, Komaki R, Mohan R. Dose and volume reduction for normal lung using intensity-modulated radiotherapy for advanced-stage non-small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2004 Mar 15;58(4):1258-67. doi: 10.1016/j.ijrobp.2003.09.086. PMID 15001271
- [Background] Gielda BT, Marsh JC, Zusag TW, Faber LP, Liptay M, Basu S, Warren WH, Fidler MJ, Batus M, Abrams RA, Bonomi P. Split-course chemoradiotherapy for locally advanced non-small cell lung cancer: a single-institution experience of 144 patients. J Thorac Oncol. 2011 Jun;6(6):1079-86. doi: 10.1097/JTO.0b013e3182199a7c. PMID 21532501
- [Background] Li Y, Wang J, Tan L, Hui B, Ma X, Yan Y, Xue C, Shi X, Drokow EK, Ren J. Dosimetric comparison between IMRT and VMAT in irradiation for peripheral and central lung cancer. Oncol Lett. 2018 Mar;15(3):3735-3745. doi: 10.3892/ol.2018.7732. Epub 2018 Jan 4. PMID 29467890
- [Background] Spoelstra FO, Pantarotto JR, van Sornsen de Koste JR, Slotman BJ, Senan S. Role of adaptive radiotherapy during concomitant chemoradiotherapy for lung cancer: analysis of data from a prospective clinical trial. Int J Radiat Oncol Biol Phys. 2009 Nov 15;75(4):1092-7. doi: 10.1016/j.ijrobp.2008.12.027. Epub 2009 Mar 26. PMID 19327915
- [Background] Inoue A, Kunitoh H, Sekine I, Sumi M, Tokuuye K, Saijo N. Radiation pneumonitis in lung cancer patients: a retrospective study of risk factors and the long-term prognosis. Int J Radiat Oncol Biol Phys. 2001 Mar 1;49(3):649-55. doi: 10.1016/s0360-3016(00)00783-5. PMID 11172945
- [Background] Vogelius IR, Bentzen SM. A literature-based meta-analysis of clinical risk factors for development of radiation induced pneumonitis. Acta Oncol. 2012 Nov;51(8):975-83. doi: 10.3109/0284186X.2012.718093. Epub 2012 Sep 5. PMID 22950387
- [Background] Wang LP, Wang YW, Wang BZ, Sun GM, Wang XY, Xu JL. Expression of interleukin-17A in lung tissues of irradiated mice and the influence of dexamethasone. ScientificWorldJournal. 2014 Mar 12;2014:251067. doi: 10.1155/2014/251067. eCollection 2014. PMID 24744681
- [Background] Kim S, Oh IJ, Park SY, Song JH, Seon HJ, Kim YH, Yoon SH, Yu JY, Lee BR, Kim KS, Kim YC. Corticosteroid therapy against treatment-related pulmonary toxicities in patients with lung cancer. J Thorac Dis. 2014 Sep;6(9):1209-17. doi: 10.3978/j.issn.2072-1439.2014.07.16. PMID 25276362
- [Background] Guilhem A, Celton B, Terminet A, Pavio C, Raschilas F, Blain H. [Radiation pneumonitis: a rare and potentially severe pneumonia. Usefulness of corticosteroids]. Rev Med Interne. 2010 Aug;31(8):e10-2. doi: 10.1016/j.revmed.2009.08.011. Epub 2010 Apr 21. French. PMID 20413191
- [Background] Sekine I, Sumi M, Ito Y, Nokihara H, Yamamoto N, Kunitoh H, Ohe Y, Kodama T, Saijo N, Tamura T. Retrospective analysis of steroid therapy for radiation-induced lung injury in lung cancer patients. Radiother Oncol. 2006 Jul;80(1):93-7. doi: 10.1016/j.radonc.2006.06.007. Epub 2006 Jul 3. PMID 16820236